CLINICAL TRIAL: NCT02350452
Title: The Impact on Ovarian Reserve of Diode Laser vs Bipolar Coagulation of Inner Lining of Ovarian Endometriomas After Laparoscopic Cystectomy: a Randomized Clinical Trial.
Brief Title: Impact on Ovarian Reserve of Diode Laser vs Bipolar Coagulation of Endometriomas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cagliari (Other)
Collaborators: University of Foggia (Other)
Responsible Party: Principal Investigator, Stefano Angioni, Associate Professor, University of Cagliari
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ENDOLASER01
Record Dates: First submitted 2015-01-19; First posted 2015-01-29 (Estimated); Last update posted 2016-04-22 (Estimated); Status verified 2016-04

CONDITIONS: Ovarian Endometrioma
Keywords: laparoscopic surgery; diode laser; AMH; AFC
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diode laser coagulation (Experimental): Diode laser coagulation of inner lining of ovarian endometrioma after laparoscopic cystectomy
  Interventions: Procedure: Diode laser coagulation
- Bipolar coaugulation (Active Comparator): Bipolar coagulation of inner lining of ovarian endometrioma after laparoscopic cystectomy
  Interventions: Procedure: Bipolar coagulation

INTERVENTIONS:
Procedure: Diode laser coagulation — Diode laser coagulation of inner lining of ovarian endometrioma after laparoscopic cystectomy
  Arms: Diode laser coagulation
Procedure: Bipolar coagulation — Bipolar coagulation of inner lining of ovarian endometrioma after laparoscopic cystectomy
  Arms: Bipolar coaugulation

SUMMARY:
Endometriosis is a benign chronic gynaecological disease that affects 10% of women of reproductive age and takes 40% of them to assisted reproduction techniques.

The purpose of the study is to compare the antimüllerian marker (AMH) and antral follicular count (AFC) , with the most common serological markers of ovarian reserve. The investigators intend to confirm their clinical utility in the assessment of ovarian function, and to promote their use in predicting decreased ovarian reserve.

The work therefore moreover arises the objective to validate the bibliographic data about using the laser for haemostasis after stripping endometriomas, to amplify knowledge available in the literature on the surgical treatment of ovarian endometriomas and on the diode laser application in minimally invasive surgery, appraising the trend of AFC and AMH levels and the possible surgical implications on fertility .

ELIGIBILITY:
Inclusion Criteria:

* regular menstrual cycles
* unilateral endometrioma greater than 35 mm
* no gynecological surgery 3-6 months before surgery
* no hormonal therapy 1 month before surgery

Exclusion Criteria:

* previous surgery for endometriosis
* hormone therapy in the month before the current surgery
* coagulation disorders
* ongoing pregnancy
* pelvic inflammatory disease
* malignant disorders
* cysts otherwise
* Gonadotropin-releasing hormone analogues or contraceptive therapy during the follow-up
* BMI≥ 30 kg/m2
* endocrinological disorders
* unable or unwilling to give written consent

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2015-01; Primary Completion 2015-08 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Anti-Müllerian hormone (AMH) serum levels | Change from AMH serum levels at 3 months after surgery

SECONDARY OUTCOMES:
Antral follicular count (AFC) | Change from AFC at 3 months after surgery, during early follicular phase

CONTACTS AND LOCATIONS:
Locations (1):
- University of Cagliari,Obstetrics and Gynecological Department,, Monserrato, Cagliari, Italy